CLINICAL TRIAL: NCT00722930
Title: Consolidation Treatment With Y90-Ibritumomab Tiuxetan In Patients With High-Risk Follicular Lymphoma With Either Partial Or Complete Response To R-Chop Induction Chemotherapy
Brief Title: Consolidation Treatment With Y90-Ibritumomab Tiuxetan After R-CHOP Induction in High Risk Patients According to Follicular Lymphoma International Prognostic Index (FLIPI) With Follicular Lymphoma
Acronym: GOTEL-FL1LC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Oncológico para el Tratamiento y el Estudio de los Linfomas (Other)
Responsible Party: Dr. Mariano Provencio, Clínica Puerta de Hierro, Servicio de Oncología Médica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOTEL-FL1LC-0701; Eudra-CT 2007-003091-19
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Follicular Lymphoma
Keywords: Follicular Lymphoma; High-risk FLIPI; R-CHOP; GOTEL; Partial; Complete; Response; Induction; Chemotherapy
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1. Consolidation with Y90 Ibritumomab Tiuxetan (Experimental): 1. Consolidation with Y90 Ibritumomab Tiuxetan
  Interventions: Drug: Y90 Ibritumomab Tiuxetan

INTERVENTIONS:
Drug: Y90 Ibritumomab Tiuxetan — Consolidation with Y90 Ibritumomab Tiuxetan

SUMMARY:
To evaluate the complete clinical response rate according to the International Working Group criteria with a consolidation treatment with 90Y-ibritumomab tiuxetan (Zevalin®) in patients with high-risk follicular lymphoma with either partial or complete response to R-CHOP induction chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Signature of the written informed consent by the subject or his/her legal representative before initiation of any trial specific procedure.
* Patients older than 18.
* Histologic diagnosis of CD20+, grade 1-3a follicular lymphoma as per the WHO classification.
* High-risk patients according to FLIPI before initiation of induction chemotherapy.
* Stage II-IV prior to initiation of induction treatment, or any stage in patients with grade 3 follicular lymphoma.
* Complete or partial response to the induction scheme.
* ECOG scale performance status 0 - 2.
* Life expectancy greater than 3 months.
* In women of childbearing age, use of a reliable contraceptive method.
* A suitable bone marrow reserve:

  * Lower than 25% Bone marrow infiltration by lymphoma.
  * Hb 10 g/dL. PMN leukocytes 1,500 cel/mm3, platelets 100,000/mm3
  * Suitable hepatic, renal and cardiac function:

    * creatinine <2,5 x UNL (upper normality limit).
    * bilirubin or ALT/AST < 2,5 x UNL

Exclusion Criteria:

* Patients with no objective clinical response to induction chemotherapy.
* > 25% bone marrow infiltration following induction chemotherapy.
* Platelets < 100,000 before radioimmunotherapy.
* Severe and/or uncontrolled concomitant disease:
* Hepatic, renal, cardiovascular, neurological or metabolic disease.
* Cardiac failure, ischemic cardiopathy, ischemic cardiopathy with a history of myocardial infarction or angor, or major ventricular arrhythmia.
* Positive regarding HBV, HCV, HIV.
* Active acute or chronic infection.
* Social, psychic or geographic disability to satisfy any of the treatment schemes.
* Pregnant and/or breastfeeding women, or adult patients of childbearing age who are not using a safe birth control device throughout the study treatment and at least 12 months thereafter.
* Known or suspected hypersensitivity, or confirmed or suspected adverse reaction to the study drugs and other related compounds (Rituximab, Ibritumomab tiuxetan, a history of sensitivity to murine proteins, dexametasone, cyclophosphamide and other anthracyclines, cytarabine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
CT scan of cervical spine, chest, abdomen and pelvis, Peripheral blood and bone marrow PCR to determine Minimal Residual Disease | 12 weeks after consolidation, then repeated every 3 months over the first 2 years, and every 6 months thereafter

SECONDARY OUTCOMES:
Objective clinical response rate (complete + partial). | 3 months
Response conversion rate | 3 months
Incidence of complete molecular responses | 3 months
Response duration | 36 months
Event-free survival. | 36 months
Progression-free survival | 36 months
Time to salvage therapy | 36 months
Lymphoma-free or specific cause-free survival | 36 months
Overall survival | 60 months
Toxicity profile and safety of the consolidation | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Principal Investigator — Clínica Puerta de Hierro
Locations (11):
- Spain (11):
  - Hospital Virgen de las Nieves, Granada, Granada
  - Clinia Puerta de Hierro, Madrid, Madrid
  - Clínica Ruber Internacional, Madrid, Madrid
  - Hospital Virgen de la Victoria, Málaga, Malaga
  - Complejo Hospitalario de Pontevedra, Pontevedra, Pontevedra
  - Instituto Oncológico San Sebastián, Donostia / San Sebastian, San Sebastián
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Sant Joan de Reus, Reus, Tarragona
  - Hospital Virgen de la Salud de Toledo, Toledo, Toledo
  - Hospital Universitario La Fe, Valencia, Valencia